CLINICAL TRIAL: NCT04460222
Title: Rotational Thromboelastometry Guided Blood Component Use in Children With Cirrhosis Undergoing Invasive Procedures: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-26
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2021-06

CONDITIONS: Cirrhosis, Liver
Keywords: ROTEM; Transfusion; Pre invasive procedure; Coagulation disorders; Pediatric liver disease
MeSH Terms: conditions — Liver Cirrhosis; Hemostatic Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotational Thromboelastometry (ROTEM) (Experimental): To prevent bleeding during invasive procedure, cirrhotic children in the ROTEM group will receive prophylactic transfusion based on the following protocol:- EXTEM CT > 80 sec - FFP will be transfused at 15 ml/kg MCF < 35 mm- Platelet will be transfused at 10 ml/kg FIBTEM MCF < 7 mm- Cryoprecipitate will be transfused at 5 ml/kg
  Interventions: Procedure: Rotational Thromboelastometry to guide blood product transfusion pre invasive procedure
- Conventional Transfusion (Active Comparator): To prevent bleeding during the procedure, cirrhotic children in the conventional group will receive prophylactic transfusion if either FFP, Platelet or Cryoprecipitate is deranged based on the following protocol
  * If INR: 1.5 - 2.5 FFP will be transfused at 10 ml/kg
  * If Platelet Count is 20,000/mm3-50,000/mm3 Platelet will be transfused at 10 ml/kg
  * If Fibrinogen < 80 mg/dl Cryoprecipitate will be transfused at 5 ml/kg
  Interventions: Procedure: Conventional transfusion methods to guide blood product transfusion pre invasive procedure

INTERVENTIONS:
Procedure: Rotational Thromboelastometry to guide blood product transfusion pre invasive procedure — Rotational Thromboelastometry will be performed pre procedure and blood component will be transfused if
  * EXTEM CT more than 80 sec then FFP will be transfused at 15 ml/kg MCF less than 35 mm then Platelet will be transfused at 10 ml/kg
  * FIBTEM MCF less than 7 mm then Cryoprecipitate will be transfused at 5 ml/kg
  Arms: Rotational Thromboelastometry (ROTEM)
Procedure: Conventional transfusion methods to guide blood product transfusion pre invasive procedure — Transfusion will be given If INR: 1.5 - 2.5 FFP will be transfused at 10 ml/kg If Platelet Count is 20,000/mm3-50,000/mm3 Platelet will be transfused at 10 ml/kg If Fibrinogen < 80 mg/dl Cryoprecipitate will be transfused at 5 ml/kg
  Arms: Conventional Transfusion

SUMMARY:
Blood products are commonly used before invasive procedures in patients with end-stage liver diseases despite cirrhosis being a thrombophilic state. Traditional coagulation tests [namely International Normalised Ratio (INR) and Platelets count] are known to be unreliable in predicting bleeding risk before invasive procedures and in representing the real coagulation status of cirrhotic patients. Notwithstanding they are still used to guide blood products administration before invasive procedures. Rotational Thromboelastometry ( ROTEM) has been shown to be effective in detecting signs of hypo-hypercoagulability possibly being an alternative method to guide blood products transfusion. The aim of this randomized controlled study is to evaluate the efficacy of ROTEM as a guide for blood products transfusion in cirrhotic children undergoing invasive procedures.

DETAILED DESCRIPTION:
Children with cirrhosis listed for invasive procedures and with deranged INR or deranged platelet count will be included in the study and will be block randomized into two groups. To prevent bleeding during the procedure, one group will receive prophylactic transfusion of either fresh frozen plasma (FFP),Platelet or Cryoprecipitate based on the values of INR, platelet and fibrinogen.The second group will undergo ROTEM based correction.

Following correction, the procedure will be done in both the groups. Patients randomized in the ROTEM group will undergo repeat ROTEM and INR, Platelet, Fibrinogen testing (depending on the component transfused), post the procedure, to look at the correction achieved. Similarly, patients randomized in the conventional group will undergo repeat INR, Platelet, fibrinogen testing depending on the component transfused.

Patients will be followed for 24 hours indoors for any evidence of bleeding or transfusion reaction.

ELIGIBILITY:
Inclusion Criteria:

•Children less than 18 years of age with histologic or image proven liver cirrhosis of any etiology with INR ≥ 1.5- ≤ 2.5 and/or Platelet count 20,000/mm3- 50,000/mm3 and who are listed for the following invasive procedures : Low risk of bleeding

1. Central venous cannulation
2. Haemodialysis catheter
3. Ascitic or Pleural tapping
4. Endoscopic variceal ligation (EVL)
5. Endoscopic sclerotherapy (EST)

High risk of bleeding 6. TIPPS 7. Endoscopic retrograde cholangiopancreatography (ERCP) with sphicterotomy 8. Percutaneous drain (PCD) Insertion 9. Biopsies other than liver biopsy

For children less than 18 years with liver cirrhosis and with a platelet count between 40,000-60,000/mm3 and INR between 1.5-2.0 who are listed for

1) Liver biopsy

Exclusion Criteria:

* Anti platelet or anti coagulant therapy in the previous 7 days
* Patients with clinical evidence of Disseminated intravascular coagulation (DIC) and/or active bleeding
* Hemodialysis in the past 7 days

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Comparison in the amount of blood products transfused between the groups | 24 hours
  To compare the amount of total component transfused (ml/kg) in Rotational Thromboelastometry guided therapy versus Conventional therapy for invasive procedures in children with cirrhosis

SECONDARY OUTCOMES:
Comparison in the amount of FFP transfused between the groups | 24 hours
  To compare the amount of FFP (ml/kg) transfused in Rotational Thromboelastometry guided therapy versus Conventional therapy for invasive procedures in children with cirrhosis
Comparison in the amount of Platelet transfused between the groups | 24 hours
  To compare the amount of Platelet transfused in Rotational Thromboelastometry guided therapy versus Conventional therapy for invasive procedures in children with cirrhosis
Comparison in the amount of Cryoprecipitate transfused between the groups | 24 hours
  To compare the amount of Cryoprecipitate transfused in Rotational Thromboelastometry guided therapy versus Conventional therapy for invasive procedures in children with cirrhosis
Post-procedure bleeding | 24 hours
  Comparison of the number of patients having bleeding episodes after procedure between the study groups
Transfusion related side effects | 5 days
  - To compare the rate of transfusion reactions in Rotational Thromboelastometry guided therapy versus Conventional therapy for invasive procedures in children with cirrhosis
Comparison between blood products costs between groups | 24 hours
  To compare the cost of transfusion components incurred in Rotational Thromboelastometry guided therapy versus Conventional therapy for invasive procedures in children with cirrhosis

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maria A, Lal BB, Khanna R, Sood V, Mukund A, Bajpai M, Alam S. Rotational thromboelastometry-guided blood component use in cirrhotic children undergoing invasive procedures: Randomized controlled trial. Liver Int. 2022 Nov;42(11):2492-2500. doi: 10.1111/liv.15398. Epub 2022 Aug 25. PMID 35977053